CLINICAL TRIAL: NCT03424070
Title: Effect of a Shoulder Roll on the Glottic View in Infants
Brief Title: Glottic View in Infants With a Shoulder Roll
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Jerrold Lerman, Clinical Professor of Anesthesiology, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Infant Shoulder Roll
Record Dates: First submitted 2017-10-17; First posted 2018-02-06 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Intubation;Difficult
Keywords: laryngoscopy; pediatric; airway; gel roll; larynx; glottis
MeSH Terms: conditions — Laryngeal Diseases

STUDY DESIGN:
Intervention Model Description: All children will undergo laryngoscopy with and without a shoulder roll (randomly assigned) during which photos will be taken of the larynx. The views will be compared using the POGO scale. Contemporaneously, the anesthesiologist's height from the table top to the lateral canthus of left eye.
Who Masked: Outcomes Assessor
Masking Description: The evaluator who measures the height between the lateral canthus of the eye of the anesthesiologist to the table top will be blinded to the presence of a shoulder roll. The evaluator who will review the final photos of the laryngeal inlet will be blinded to the order of the positioning.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laryngoscopy view with a shoulder roll (Active Comparator): The primary outcome is the difference in the height of the lateral canthus of the eyelid of the laryngoscopist above the OR table during laryngoscopy with and then without the shoulder roll. These two positions will be compared using photos of the best glottic view taken during laryngoscopy with a shoulder roll in place. Then a photo of the best glottic view will be taken during laryngoscopy without the shoulder roll in place. These two views will be compared by a blinded anesthesiologist using the POGO scale.
  Interventions: Other: Shoulder Roll
- Laryngoscopy without a shoulder roll (Placebo Comparator): The primary outcome is the difference in the height of the lateral canthus of the eyelid of the laryngoscopist above the OR table during laryngoscopy without and then with the shoulder roll. These two positions will be compared using photos of the best glottic view taken during laryngoscopy with a shoulder roll in place. Then a photo of the best glottic view will be taken during laryngoscopy without the shoulder roll in place. These two views will be compared by a blinded anesthesiologist using the POGO scale.
  Interventions: Other: No shoulder roll (placebo)

INTERVENTIONS:
Other: Shoulder Roll — The POGO score assesses the percent of the glottic opening that can be seen with and without the shoulder roll.
  Other Names: jelly roll
  Arms: Laryngoscopy view with a shoulder roll
Other: No shoulder roll (placebo) — Placebo
  Arms: Laryngoscopy without a shoulder roll

SUMMARY:
This study compares the distance from the operating table to the eye of the laryngoscopist while intubating the trachea with or without a shoulder roll. A photo of the glottic opening will compare the glottic views in both positions.

DETAILED DESCRIPTION:
On the day of the surgery, healthy infants will be evaluated by an anesthesiologist for a preoperative clearance and suitability for inclusion in the study. If the infants are eligible, the parents will receive a detailed explanation of the study that is written into the consent form. Written consent will be obtained from those parents who are willing to enroll their children in the study. After consent, the concealed randomization code for the next subject in the study will be opened to determine the sequence of the positioning as described below.

The infants will be unpremedicated. In the operating room, anesthesia will be induced using a standard inhalational induction (that includes, 70 % nitrous oxide and 30 % oxygen followed by 8% sevoflurane). Upon the loss of eyelash reflex, ventilation will be assisted and intravascular (IV) access will be secured. Once IV access is established, Propofol, 3 mg/kg will be administered and the lungs ventilated with 8% sevoflurane in 100% oxygen for 1 minute. The randomization code will then determine the order of the laryngoscopy: either no shoulder roll or a 2 inch shoulder roll first, then the alternative position. For both positions, direct laryngoscopy using a #1 size straight Miller blade will expose the larynx to obtain the optimal glottic view. At this point, the distance from the lateral canthus of the eye of the anesthesiologist to the level of the table will be recorded (distance A) using a standard measure anchored on the operating room table top and a photo of the glottic opening will be taken using a high-quality digital hand-held camera. This photo will be referred to as photo 1. The shoulder roll will either be removed or inserted under the shoulders (based on the randomization) while the anesthesiologist holds the laryngoscopic view of the larynx. The anesthesiologist's head will then move (if necessary) up or down to establish the optimal view of the larynx again and the distance from the lateral canthus of the eye of the anesthesiologist to the table top will again be measured (distance B). A photo of the laryngoscopy view (photo 2) will be taken. The entire laryngoscopy will take less than 30 seconds. If the child desaturates to less than 93%, the study will be aborted and the lungs ventilated. An anesthesiologist, who is blind to the study hypothesis, will evaluate the photos of the glottis view the Percent of Glottic Opening scale (POGO) in 10% increments. The primary outcome will be the distance from the lateral canthus of the anesthesiologist's eye to the level of the table with and without a shoulder roll (distance A and distance B) will be compared using paired t-test. (P<0.05 will be accepted). The secondary outcome will be the glottic views (photos 1 and picture 2) compared using the Kruskall Wallis test.

ELIGIBILITY:
Inclusion Criteria:

* 0-12 months of age
* American Society of Anesthesiologists (ASA) I-II
* Elective non-airway surgery under general anesthesia

Exclusion Criteria:

* Emergency surgeries
* Patients in whom difficult airway is expected
* Obese patients in whom BMI >95 percentile for age
* Patients with untreated gastroesophageal reflux
* Full stomach patients

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-02-18 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
The height from the anesthesiologist's (cm) eye to the table top with and without a shoulder roll | One day
  Height in centimeters from the lateral canthus of the eye of the anesthesiologist to the table top.

SECONDARY OUTCOMES:
The view of the glottic opening (in percent) with and without a shoulder roll | 1 day
  The view of glottic opening with and without a shoulder roll (secondary outcome) will be compared in photos and measured as a percent of the full length of normal vocal cords (from a standard photograph)

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold Lerman, Principal Investigator — Women & Children's Hospital/ Great Lakes Anesthesiology
Locations (1):
- Women and Children's Hospital of Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenland KB, Edwards MJ, Hutton NJ, Challis VJ, Irwin MG, Sleigh JW. Changes in airway configuration with different head and neck positions using magnetic resonance imaging of normal airways: a new concept with possible clinical applications. Br J Anaesth. 2010 Nov;105(5):683-90. doi: 10.1093/bja/aeq239. Epub 2010 Sep 15. PMID 20846964
- [Background] Kim EH, Ji SH, Song IK, Lee JH, Kim JT, Kim HS. Simple method for obtaining the optimal laryngoscopic view in children: A prospective observational study. Am J Emerg Med. 2017 Jun;35(6):867-870. doi: 10.1016/j.ajem.2017.01.048. Epub 2017 Jan 24. PMID 28139308
- [Background] Black AE, Flynn PE, Smith HL, Thomas ML, Wilkinson KA; Association of Pediatric Anaesthetists of Great Britain and Ireland. Development of a guideline for the management of the unanticipated difficult airway in pediatric practice. Paediatr Anaesth. 2015 Apr;25(4):346-62. doi: 10.1111/pan.12615. Epub 2015 Feb 16. PMID 25684039
- [Derived] Alfahel W, Gopinath A, Arheart KL, Gensler T, Lerman J. The Effects of a Shoulder Roll During Laryngoscopy in Infants: A Randomized, Single-Blinded, Crossover Study. Anesth Analg. 2020 Oct;131(4):1210-1216. doi: 10.1213/ANE.0000000000004802. PMID 32925342